CLINICAL TRIAL: NCT02256527
Title: REWARDS-Premier TLX (Registry Experience at the WAshington Hospital CenteR, DeS - Premier Taxus-Liberte vs Xience V)
Brief Title: REWARDS Premier Taxus-Liberte vs Xience V
Status: Completed | Type: Observational
Sponsor: Medstar Health Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: REWARDS Premier TLX
Record Dates: First submitted 2014-10-01; First posted 2014-10-03 (Estimated); Last update posted 2016-07-14 (Estimated); Status verified 2016-07

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Promus Premier: observational data
  Interventions: Other: Observational

INTERVENTIONS:
Other: Observational — compare data

SUMMARY:
Multicenter, retrospective registry to collect baseline, clinical, procedural, in hospital and 9-12 month follow-up data to compare major adverse cardiac events in patients receiving Promus Premier drug eluting stent to data already collected from the REWARDS-TLX Registry in which patients received either the Taxus Liberte or XIENCE V drug eluting stent.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years of age or older
* Underwent PCI with Promus Premier (alone) DES

Exclusion Criteria:

* Underwent PCI with a non-Promus Premier DES during the same index procedure
* Patients not taking, or unable to take, dual antiplatelet therapy (aspirin plus clopidogrel, prasugrel, or ticagrelor)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients male or female, 18 years or older who have undergone percutaneous coronary intervention with Promus Premier (alone) drug eluting stent
Sampling Method: Non-Probability Sample
Enrollment: 917 (Actual)
Dates: Start 2014-09; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Major adverse cardiac event | 1 year
  composite of all-cause death, Q-wave myocardial infarction, and target vessel revascularization

CONTACTS AND LOCATIONS:
Locations (1):
- Washington Hospital Center, Washington D.C., District of Columbia, United States